CLINICAL TRIAL: NCT06347796
Title: Chronic Subdural Hematoma Treatment With Embolization Versus Surgery Study
Acronym: CHESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0160; UG3NS128397 (NIH); UH3NS128397 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma (CSDH); middle meningeal artery embolization (MMAE)
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Middle Menningeal Artery Embolization (MMAE) (Experimental)
  Interventions: Device: Middle Meningeal Artery Embolization (MMAE)
- Conventional Surgery (Craniotomy or Burr Holes) (Active Comparator)
  Interventions: Procedure: Conventional Surgery

INTERVENTIONS:
Procedure: Conventional Surgery — Conventional surgery is surgical drainage through burr holes or craniotomy.
  Arms: Conventional Surgery (Craniotomy or Burr Holes)
Device: Middle Meningeal Artery Embolization (MMAE) — Particle embolization of the middle meningeal artery with micron variants of the Embosphere Microspheres or CONTOUR Embolization Particles device.
  Arms: Middle Menningeal Artery Embolization (MMAE)

SUMMARY:
The goal of this clinical trial is to test in moderately symptomatic chronic subdural hematoma (CSDH) patients if middle meningeal artery embolization (MMAE) can be used as an alternative to conventional open surgery. The main questions it aims to answer are:

* Compared to open conventional surgery, does MMAE reduce the need for rescue surgery or deaths?
* What is the safety of MMAE and conventional open surgery in these patients?

Participants will be asked to:

* Share their medical history and undergo physical examinations
* Have blood drawn
* Have CT scans of the head
* Answer questionnaires
* Undergo MMAE or conventional open surgery
* Provide information about possible adverse events Researchers will compare participants in the MMAE group with those in the conventional open surgery group to see if there is a reduced need for rescue surgery or deaths and evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-90 years inclusively.
2. Per CT of the head, (one of the following): Unilateral convexity CSDH measuring at least 10 mm in thickness OR Bilateral CSDH if only one side is considered for treatment and the contralateral side is asymptomatic and < 5 mm in thickness.
3. CSDH at least 2/3 isodense or hypodense, verified on axial CT slice used to measure the thickness of the qualifying CSDH.
4. Qualifying baseline head CT performed within the 7 days prior to randomization.
5. Able to undergo assigned treatment within 72 hours after randomization.
6. Patient or legally authorized representative agrees to be randomized, and provides written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

1. Secondary cause apart from trauma for the qualifying SDH, such as an underlying vascular abnormality or tumor.
2. Tentorial or interhemispheric SDH.
3. Secondary to CSDH, MRC of 0, 1, 2, or 3 in any muscle group contralateral to the side of the CSDH 4.
4. Pre CSDH mRS of 5 or higher.
5. Secondary to CSDH, patient is unable to complete TUG (i.e.,TUG > 120 seconds, unable to walk, or tries TUG but quits in ≤ 120 seconds). Note: This criterion does not apply if the patient does not complete TUG for reason other than CSDH.
6. Secondary to CSDH, ASR of 0, 1, or 2.
7. Emergent surgical evacuation such as open craniotomy, burr hole drainage, or Subdural Evacuating Port System (SEPS) is required for the patient.
8. Unable to withhold all antiplatelet agents or OACs for the first 7 days after randomization.
9. Indication that withdrawal of care will be implemented for the qualifying SDH.
10. Prior surgical treatment for CSDH if the surgery is less than 30 days prior to randomization.
11. On tranexamic acid.
12. Platelet count of <100,000 per microliter refractory to transfusion.
13. Coagulopathy that cannot be corrected to an INR of ≤1.5.
14. Known contraindications to angiography.
15. Known intolerance to occlusion procedures.
16. Known vascular anatomy (small artery size) or blood flow (high vascular resistance peripheral to the feeding arteries) that precludes catheter placement or embolic agent (Embosphere Microspheres or CONTOUR particles) injection.
17. Known presence of collateral vessel pathways potentially endangering normal territories or cranial nerves during embolization.
18. Known large diameter arteriovenous shunt, i.e., where the blood does not pass through an arterial/capillary/venous transition but directly from an artery to a vein or presence of patent extra-to-intracranial anastomoses (where study embolization devices could pass directly into the internal carotid artery, vertebral artery, or intracranial vasculature) that cannot be addressed with coil embolization.
19. Patient has a known active systemic infection or sepsis.
20. Patient is pregnant, planning to become pregnant, or lactating.
21. Life expectancy of less than 6 months due to comorbid terminal conditions.
22. Concurrent participation in another research protocol for investigation of an experimental therapy.
23. Known or suspected to not be able to comply with the study protocol.
24. No measurable deficit secondary to the CSDH on the Timed Up and Go [TUG], Aphasia Severity Rating [ASR], or MRC. At baseline, a measurable deficit on the TUG is defined as: time >10 seconds. At baseline, a measurable deficit on the ASR is defined as: a score<4. At baseline, a measurable deficit on the MRC is defined as: a score < 5 in any muscle group contralateral to the site of the CSDH.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Need for Rescue Surgery or Death | Within 180-210 days of randomization
  Participants who need rescue surgery or die.

SECONDARY OUTCOMES:
Safety of MMAE and Conventional Open Surgery | Within 180 days of randomization.
  The proportion of subjects with symptomatic ischemic stroke, serious/life threatening adverse events, worsening of neurological status (a decline of 1 point on the Markwalder scale) or development of new disabling neurological symptoms, seizures, and/or cranial neuropathy.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri Healthcare, Columbia, Missouri
  - Washington University, St. Louis, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - JFK Neuroscience Institute, JFK University Medical Center, Edison, New Jersey
  - Rutgers, The State University of New Jersey, Newark, New Jersey
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University of Pennyslvania, Philadelphia, Pennsylvania
  - Philadelphia Neurological Institute, Upland, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center-Houston, Houston, Texas
  - University of Texas Health Science Center-San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No